CLINICAL TRIAL: NCT01346033
Title: An Evaluation of a Non-invasive Diabetes Screening Device in Subjects With Type 2 Diabetes
Brief Title: Evaluation of SCOUT DS in Subjects With Type 2 Diabetes
Acronym: TCOYD
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2714
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Adults 18 years and older; Taking Control of Your Diabetes Health Fair
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Those with Type 2 diabetes: All subjects have been diagnosed with type 2 diabetes.

SUMMARY:
The primary objective of the trial is to collect SCOUT DS and Hemoglobin A1c measurements of subjects who have been diagnosed with Type 2 diabetes.

DETAILED DESCRIPTION:
Previous studies have excluded subjects with Type 2 diabetes. The primary objective of this study is to correct an imbalance in the disease prevalence of the data set used to develop the SCOUT DS diabetes screening algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Self-reported diagnosis of type 2 diabetes

Exclusion Criteria:

* Not diagnosed with type 2 diabetes

  * Diagnosed with type 1 diabetes
  * Known to be pregnant (Self Reported)
  * Receiving dialysis or having known renal compromise
  * Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
  * Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Attendees of the Taking Control of Your Diabetes Health Fair, San Diego CA Convention Center
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Validation of SCOUT DS algorithm for detecting known type 2 diabetes | 1 day
  Collect SCOUT DS and Hemoglobin A1c measurements of subjects with Type 2 Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Kabongo, MD,PhD, Principal Investigator — Accelovance San Diego
Locations (1):
- San Diego Convention Center, San Diego, California, United States